CLINICAL TRIAL: NCT00063115
Title: Event-Related fMRI Analysis of Patients With Ideomotor Apraxia During Transitive and Intransitive Hand Gesturing
Brief Title: Using fMRI to Understand the Roles of Brain Areas for Fine Hand Movements
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030230; 03-N-0230
Record Dates: First submitted 2003-06-19; First posted 2003-06-20 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-07-02

CONDITIONS: Ideomotor Apraxia
Keywords: Praxis Movements; Pantomime; Statistical Parametric Mapping; Functional Connectivity; Path Analysis; Ideomotor Apraxia; Healthy Volunteer; HV
MeSH Terms: conditions — Apraxia, Ideomotor

SUMMARY:
Ideomotor apraxia, a disorder that affects patients with stroke and a variety of other brain lesions, features disturbed timing, sequence, and spatial organization of skilled movements. This study will look at how different areas of the human brain control fine hand movements.

Thirty-five participants 21 years and older will be enrolled in this study-25 healthy, right-handed people, and 10 stroke patients. They will undergo two outpatient sessions, each lasting up to 3 hours. The first visit for the stroke patients will occur between 2 weeks and 3 months after the stroke; the second visit will be at least 6 months after the stroke.

Participants will have a physical exam, give a medical history, and complete a questionnaire. Then they will undergo magnetic resonance imaging (MRI) scans. They will lie in the MRI scanner and will be asked to do a number of skilled hand movements using the right hand (such as pretending to use a hammer or waving goodbye) in response to directions that will appear on a screen mounted over their head. Their movements will be recorded on videotape during the procedures.

DETAILED DESCRIPTION:
OBJECTIVE: The present study focuses on evaluating neural activation patterns underlying praxis movements in normal controls and in patients with ideomotor apraxia using event-related functional magnetic resonance imaging (fMRI). Ideomotor apraxia is a disorder affecting patients with stroke and a variety of other brain lesions. The disorder involves disturbed timing, sequence, and spatial organization of skilled movements, during the execution and probably also preparatory phases. As a consequence, patients suffer from incorrect temporal and spatial components to movements as evidenced during pantomime of transitive (object/tool related) and intransitive (independent of object/tool use) gestures. Thus far, damage to posterior parietal regions and parietofrontal circuits has been implicated in significantly contributing to this disorder. However, little is known about the mechanism of cortical reorganization following damage, notably during recovery process. We hypothesize that recruitment of parallel and contralateral motor pathways compensates for reduced communication within parietofrontal circuits which prevents accurate motor performance.

STUDY POPULATION: We will study two groups of participants: one group of patients with ideomotor apraxia and one group of healthy subjects.

DESIGN: We will measure fMRI activation on transitive and intransitive gestures in 10 patients with ideomotor apraxia during subacute and chronic stage compared to 25 normal controls. The design of the behavioral paradigm incorporates a distinct period of planning prior to each movement.

OUTCOME MEASURES: The design of this study allows evaluating any differences in the planning and execution phases between patients and controls. Further analysis will examine patterns of functional connectivity between activated brain areas, notably their altered interactions in ideomotor apraxia. Of special interest is the putative engagement of perilesional or even remote brain areas in a neuronal network during attempted recovery from motor deficit.

It is expected from the study that a better understanding of cortical plasticity compensating for motor deficits in ideomotor apraxia can be therapeutically exploited, notably in the rehabilitation process.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers.

Patients diagnosed with ideomotor apraxia with a single left hemisphere stroke will be included.

The lesion will be located in any part of the frontal and parietal areas or both, as well as their connections.

EXCLUSION CRITERIA:

Subjects with abnormal neurologic examinations, previous or current neurological and psychiatric disorders will be excluded.

Subjects under age 21, pregnant or mentally impaired will also be excluded.

Ideomotor apraxic patients with a second neurologic disorder including more than one brain lesion of the inability to cooperate fully will be excluded.

Patients with a history of significant medical disorders such as cancers will be excluded.

MRI experiments will not be performed in subjects or patients who have pacemakers, brain stimulators, dental implants or metallic braces, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, insulin pumps, or shrapnel fragments.

Welders and metal workers are also at risk for injury because of possible small metal fragments in the eye of which they may be unaware. Subjects will be screened for these contraindications prior to the study.

MRI experiments will not be performed on pregnant women.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35
Dates: Start 2003-06-16; Study Completion 2008-07-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Haaland KY, Harrington DL, Knight RT. Neural representations of skilled movement. Brain. 2000 Nov;123 ( Pt 11):2306-13. doi: 10.1093/brain/123.11.2306. PMID 11050030